CLINICAL TRIAL: NCT01208064
Title: Double Blind Randomized Phase III Study of Maintenance Pazopanib Versus Placebo in NSCLC Patients Non Progressive After First Line Chemotherapy. MAPPING, an EORTC Lung Group Study.
Brief Title: Pazopanib Hydrochloride or a Placebo in Treating Patients With Non-Small Cell Lung Cancer Who Have Received First-Line Chemotherapy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: based on IDMC decision
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EORTC-08092; 2010-018566-23 (EudraCT Number); EU-21072
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pazopanib (Experimental): 2 weeks at 600mg and then maintenance at 800mg
  Interventions: Drug: pazopanib hydrochloride; Other: laboratory biomarker analysis; Other: pharmacogenomic studies; Other: pharmacological study; Procedure: quality-of-life assessment
- Placebo (Placebo Comparator): placebo match 2 weeks at 600mg and then maintenance at 800mg
  Interventions: Other: laboratory biomarker analysis; Other: pharmacogenomic studies; Other: pharmacological study; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: pazopanib hydrochloride
  Arms: Pazopanib
Other: laboratory biomarker analysis
Other: pharmacogenomic studies
Other: pharmacological study
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether pazopanib hydrochloride is more effective than a placebo in treating patients with non-small cell lung cancer that has not progressed after first-line chemotherapy.

PURPOSE: This randomized phase II/III trial is studying how well giving pazopanib hydrochloride works and compares it with giving a placebo in treating patients with non-small cell lung cancer who have received first-line chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the therapeutic benefit, in terms of overall survival, of maintenance pazopanib hydrochloride in patients with non-small cell lung cancer who have not progressed after first-line chemotherapy.

Secondary

* To compare progression-free survival (PFS) overall and at specific time points (6 and 12 months).
* To document the toxicity profile of pazopanib hydrochloride according to the CTCAE v 4.
* To assess the use of C-reactive protein (CRP) in the detection of progression of disease in the maintenance phase of therapy.
* To compare quality-of-life of patients on maintenance therapy.
* To compare discontinuation rate/treatment compliance of patients treated with these regimens.
* To collect health economics data on resource utilization as documented by the EQ-5D generic QoL instrument.

Tertiary (correlative)

* To evaluate the effect of germline genetic variations on drug response (pharmacogenetics) using PAX gene.
* To find relevant biomarkers of VEGFR pathways from plasma samples.
* To obtain the pharmacokinetics of pazopanib hydrochloride at 600 and 800 mg.
* To evaluate biomarkers in tumor tissue.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to center, histology (squamous vs nonsquamous), performance status (0-1 vs 2 up to 15% of patients), and response to initial chemotherapy (complete response/partial response vs stable disease). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive an oral placebo daily on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral pazopanib hydrochloride daily on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients complete quality-of life-questionnaires (QLQ-C30 and QLQ-LC13) at baseline, 6 weeks, 14 weeks, and 22 weeks.

Health economics data on resource utilization are collected and documented using the EQ-5D questionnaire.

Blood samples may be collected periodically for pharmacokinetics and pharmacogenetic studies. Samples are analyzed for germline genetic variations on drug response, relevant biomarkers of VEGFR pathways, and concentration of pazopanib hydrochloride. Previously collected tumor tissue is analyzed for biomarkers.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) meeting the following criteria:

  * Any histology
  * Stage IIIB-IV disease
* Newly diagnosed or recurrent disease (after surgery or radical radiotherapy) proven on cytology or histology before induction chemotherapy

  * In case of adjuvant chemotherapy after previous surgery, time interval from start of previous treatment to induction chemotherapy for metastatic disease is 12 months
* May or may not have measurable disease as defined by RECIST criteria
* Must not have progressed during the 4 courses of initial chemotherapy

  * For patient presenting with measurable disease, there must be documented radiographic evidence of response (complete response, partial response, or stable disease) according to RECIST 1.1 criteria
  * For patients without measurable disease, there must be no symptomatic/clinical progression
* EGFR wild-type or unknown (known EGFR mutations are not eligible)
* Brain metastases allowed provided they are controlled and the patient must present with a performance status (PS) of 0-1 after the 4 courses of chemotherapy and at least 1 week off steroids
* No known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage, including any of the following:

  * Large protruding endobronchial lesions in the main or lobar bronchi

    * Endobronchial lesions in the segmented bronchi are allowed
  * Lesions extensively infiltrating the main or lobar bronchi

    * Minor infiltrations in the wall of the bronchi are allowed
  * Lesions infiltrating major pulmonary vessels (contiguous tumor and vessels)

    * Tumors touching but not infiltrating (abutting) the vessels are acceptable

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-2

  * PS 2 capped at 15% of the study population
  * Elderly population (i.e., > 70 years old) capped at 15% and must be PS 0-1
* Life expectancy ≥ 12 weeks
* ANC ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 9 g/dL
* PT or INR ≤ 1.2 times upper limit of normal (ULN)
* PTT ≤ 1.2 times ULN
* Bilirubin ≤ 1.5 times ULN
* AST/ALT ≤ 2.5 times ULN
* Serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 50 mL/min
* Urine protein:creatinine ratio ≤ 1 OR ≤ 1.0 g of protein by 24-hour urine collection
* May only be randomized in this trial once
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception 2 weeks prior to, during, and for at least 1 month after completion of study therapy
* Corrected QT interval (QTc) ≤ 480 msec on normal 12-lead ECG

  * If QTc interval is > 480 msec, then 2 additional ECGs should be obtained over a brief period of time (e.g., within 15-20 minutes) to confirm the abnormality and the average QTc interval will be determined from the 3 ECG tracings by manual evaluation and will be used to determine if the patient will be excluded from the study
* No history of any of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
* No NYHA class III-IV congestive heart failure (no class II, III, or IV for elderly patients)
* LVEF normal
* No other malignancy within the past 2 years except for non-small cell lung cancer
* No poorly controlled hypertension, defined as blood pressure (BP) > 140/90 mm Hg

  * Initiation or adjustment of antihypertensive medications is permitted prior to study entry provided blood pressure is reassessed on two occasions that are separated by a minimum of 1 hour and the mean systolic BP/diastolic BP values must be ≤ 140/90 mm Hg
* No cerebrovascular accident (at any time in the past), transient ischemic attack, deep venous thrombosis (DVT), or pulmonary embolism within the past 6 months

  * Patients with recent DVT who have been treated with therapeutic anticoagulating agents and remained stable for at least 6 weeks are eligible
* No hemoptysis within the past 6 weeks (patients with a history of hemoptysis associated with metastatic disease must undergo a bronchoscopy to rule out endobronchial lesions and patients with an endobronchial lesion will be excluded from the study)
* No history of clinically significant gastrointestinal disorders, including any of the following:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel that could affect the absorption of the study drug
  * Active peptic ulcer disease
  * Known intraluminal metastatic lesions with risk of bleeding
  * Inflammatory bowel disease
  * Ulcerative colitis
  * Other gastrointestinal conditions with increased risk of perforation
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No evidence of active bleeding or bleeding diathesis
* No trauma within the past 28 days
* No nonhealing wound, fracture, or ulcer
* No known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib hydrochloride
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No ongoing toxicity from prior anticancer therapy that is > grade 1 (except alopecia) and/or that is progressing in severity
* At least 6 months since prior amiodarone
* At least 14 days since prior CYP3A4 substrates
* At least 2 weeks since prior palliative radiotherapy
* No major surgery within the past 28 days
* No prior multi-target tyrosine kinase inhibitor (TKI), bevacizumab, or cetuximab (as part of induction therapy)
* Prior radical radiotherapy allowed provided it was at least 12 months from start of induction chemotherapy for metastatic disease
* Concurrent anticoagulant therapy allowed provided the patient's PT, INR, or PTT is stable and within the recommended range for the desired level of anticoagulation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Progression-free survival (PFS) overall and at 6 and 12 months
Toxicity
Correlation of C-reactive protein with PFS at weeks 6, 14, and 22
Quality of life
Comparison of discontinuation rate with treatment compliance
Health economics

CONTACTS AND LOCATIONS:
Overall Officials: Mary O'Brien, MD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (22):
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Regional De La Citadelle, Liège
  - Clinique et Maternité Sainte Elisabeth, Namur
- National Cancer Institute, Cairo, Egypt
- France (2):
  - Centre Georges-Francois-Leclerc, Dijon
  - Assistance Publique - Hôpitaux de Marseille - Assistance Publique - Hôpitaux de Marseille - Hopital Nord, Marseille
- Germany (2):
  - Klinik Loewenstein, Löwenstein
  - UniversitaetsMedizin Mannheim, Mannheim
- University General Hospital Heraklion, Heraklion, Greece
- Netherlands (3):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Isala Klinieken, Zwolle
- University Clinic Golnik, Golnik, Slovenia
- United Kingdom (9):
  - Royal Marsden - Surrey, Sutton, England
  - Western General Hospital, Edinburgh
  - Guy's and St Thomas' NHS, London
  - Royal Marsden Hospital, London
  - Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Weston Park Hospital, Sheffield
  - Royal Marsden Hospital, Sutton
  - King's Mill Hospital, Sutton in Ashfield